CLINICAL TRIAL: NCT01934296
Title: Chronic Effects of Deep Brain Stimulation on Cortical Local Field Potentials in Parkinson's Disease and Dystonia
Brief Title: Chronic Effects of DBS in Parkinson's Disease and Dystonia
Acronym: Activa PC+S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Philip Starr, Professor, Neurological Surgery, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Activa PC+S
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Parkinson's Disease; Isolated Dystonia
Keywords: deep brain stimulation; cortical recording; neuroprosthesis
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chronic brain recording (Experimental): This is a one-arm, single-center study of the neurophysiology of human movement disorders with two goals: 1) Assess the feasibility of chronic brain recording using a novel fully implantable pulse generator (Medtronic Activa PC+S), which has the capability of sensing and storing local field potentials (LFPs) recorded from implanted electrodes, in addition to providing therapeutic deep brain stimulation (DBS). 2) Study acute and chronic effects of therapeutic DBS on cortical LFPs. 3) Study feasibility of the use of brain signals as feedback either directly to the patient or for DBS stimulation adjustments.
  Interventions: Device: Activa PC+S

INTERVENTIONS:
Device: Activa PC+S — Surgical implantation of Activa PC+S as one component of a therapeutic DBS system implantation

SUMMARY:
The purpose of this study is to use an investigational device to record brain activity for 12-24 months following surgical implantation of deep brain stimulation (DBS) systems. The goal of the study is better understanding of brain activity in movement disorders and how they relate to DBS, not to bring new devices to market.

ELIGIBILITY:
Inclusion Criteria(both groups):

* Ability to give informed consent for the study
* Movement disorder symptoms that are sufficiently severe, in spite of best medical therapy, to warrant surgical implantation of deep brain stimulators according to standard clinical criteria

Inclusion criteria (Isolated dystonia):

* Age 22-75
* Isolated dystonia that is generalized or segmental, that must affect one or - Stable doses of anti-dystonia medications (such as Artane, Baclofen, or Clonopin) for at least 30 days prior to baseline assessment
* For patients with craniofacial involvement, prior treatment with botulinum toxin with failure to adequately control dystonia symptoms.

Inclusion criteria (PD):

* Age 30-75
* Bilateral disease (Hoehn and Yahr stage 2 or greater)
* Has been treated with levodopa/carbidopa, and with a dopamine agonist, at the maximal tolerated doses as determined by a movement disorders neurologist
* Stable doses of antiParkinsonian medications for at least 30 days prior to their baseline assessment
* Significant disability in the setting of optimal medical management by a movement disorders neurologist. Disability may be due to tremor that is unresponsive to medications, or to motor fluctuations
* UPDRS-III score off medication between 20 and 60
* Improvement of at least 30% in the baseline UPDRS-III on medication score, compared to the baseline off-medication score.

Exclusion Criteria (both groups):

* Pregnancy or breast feeding
* MRI showing cortical atrophy out of proportion to age
* MRI showing focal brain lesions that could indicate a non-idiopathic movement disorder,
* Major comorbidity increasing the risk of surgery (prior stroke, severe hypertension, severe diabetes, or need for chronic anticoagulation other than aspirin)
* Inability to comply with study follow-up visits
* Any prior intracranial surgery
* Mood depression with a Beck depression inventory score of > 17 on baseline screening
* Significant cognitive impairment (MoCA<25).
* History of seizures
* Immunocompromised
* Has an active infection
* Requires diathermy, electroconvulsive therapy (ECT) or transcranial magnetic - Has an implanted electronic device such as a neurostimulator, cardiac pacemaker or medication pump.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-11; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Starr, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Surgical Movement Disorders Center, San Francisco, California, United States

REFERENCES:
- [Result] Swann NC, de Hemptinne C, Miocinovic S, Qasim S, Ostrem JL, Galifianakis NB, Luciano MS, Wang SS, Ziman N, Taylor R, Starr PA. Chronic multisite brain recordings from a totally implantable bidirectional neural interface: experience in 5 patients with Parkinson's disease. J Neurosurg. 2018 Feb;128(2):605-616. doi: 10.3171/2016.11.JNS161162. Epub 2017 Apr 14. PMID 28409730

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Brain Recording
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Brain Recording
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.44 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Parkinson's Disease With Reliable Cortical and Sub-cortical Brain Signals
Description: To report number of PD patients with reliable cortical and subcortical brain signal recorded using Activa PC+S.
Time Frame: 24 months
Population: 5 patients with Parkinson's disease
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Brain Recording
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: 2 years for each patient
Arm/Group | Chronic Brain Recording
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Brain Recording (N=9)
Cerebrospinal Fluid (CSF) collected under scalp (Surgical and medical procedures) | 1 (1) — One patient had a transient sterile fluid collection, consistent with CSF, under the frontal scalp postoperatively that appeared in the morning after sleep and disappeared in the upright posture.
Fatigue after surgery (Surgical and medical procedures) | 1 (1) — One patient reported fatigue after surgery concurrent with reduction in levodopa.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT01934296/Prot_SAP_000.pdf